CLINICAL TRIAL: NCT06201663
Title: Safety and Efficacy of Romiplostim in Chemotherapy-Induced Thrombocytopenia in Children and Adolescents With Solid Malignancy
Brief Title: Romiplostim in Chemotherapy-Induced Thrombocytopenia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FAMSU MD343/2023
Record Dates: First submitted 2023-12-30; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: Chemotherapy-induced Thrombocytopenia; Solid Malignancy
MeSH Terms: interventions — romiplostim

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional group (Experimental): Patients with CIT fulfilling the inclusion criteria will receive romiplostim subcutaneously weekly, either at the time of nadir of a delayed chemotherapy cycle or on the first day of the subsequent chemotherapy cycle and continue until the completion of chemotherapy for maximum 12 weeks.
  Starting dose will be 3 μg/kg with the escalation of the dose weekly by 2 μg/kg (maximum dose 10 μg/kg) when the platelet increment was less than 25 x10e9/L to maintain platelet counts above 75x10e9/L.
  Interventions: Drug: Romiplostim
- Control group (No Intervention): Patients with CIT fulfilling the inclusion criteria randomized to the control group will not receive romiplostim injections.
  Patients are allowed to received supportive care according to the standard of care protocols.

INTERVENTIONS:
Drug: Romiplostim — Weekly subcutaneous injections
  Other Names: TPO-RA
  Arms: Interventional group

SUMMARY:
Prospective interventional randomized controlled trial to assess safety and efficacy of romiplostim in chemotherapy-induced thrombocytopenia in children and adolescents with solid malignancy

DETAILED DESCRIPTION:
Chemotherapy-induced thrombocytopenia (CIT) frequently complicates cancer treatment causing delays in treatment and dose reduction for subsequent administration of cancer-directed treatment.

Romiplostim is a potential agent that can improve platelet counts, allowing the resumption of chemotherapy, decreasing the need for platelet transfusions, and increasing the nadir platelet counts thus improving dose intensity.

ELIGIBILITY:
Inclusion Criteria:

Age: 1- 18 years. Patients diagnosed with solid malignancy based on clinical, histopathological features, and /or immunohistochemical staining.

Patients with chemotherapy-induced thrombocytopenia defined as either

* severe thrombocytopenia either clinically with high bleeding score or laboratory by platelet count reaching critical level < 20x10e9/L requiring platelet transfusion at time of chemotherapy cycle nadir.
* delayed recovery of platelet count: a platelet count of less than 100 x10e9/L for 3 weeks from the first day of chemotherapy cycle administration or the previous dose was reduced by >20% due to low platelet count <100×10e9/L.

Exclusion Criteria:

* Patients with second primary neoplasm.
* Patients with relapsed/refractory solid malignancy.
* Presence of primary or metastatic liver cancer.
* History of a prior symptomatic venous thromboembolic event (VTE) or arterial ischemic events.
* Patients with thrombocytopenia due to other etiologies e.g., underlying inherited thrombocytopenia.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-17 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Hematologic response | 12 weeks
  Platelet count increase to > 75 x 10e9/L, as well as toleration of chemotherapy resumption for at least 8 weeks or two cycles without subsequent chemotherapy dose reduction or dose delay because of recurrent CIT

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Children's Hospital, Cairo, Egypt